CLINICAL TRIAL: NCT03897179
Title: INVSENSOR00032 and INVSENSOR00033 Respiration Rate Clinical Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19608
Record Dates: First submitted 2019-03-20; First posted 2019-04-01 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00032 and INVSENSOR00033 test group (Experimental): All subjects will be enrolled into the test group and will receive the INVSENSOR00032 and/or INVSENSOR00033 device.
  Interventions: Device: INVSENSOR00032 and INVSENSOR00033

INTERVENTIONS:
Device: INVSENSOR00032 and INVSENSOR00033 — Investigational pulse oximeter device

SUMMARY:
This study compares the performance of respiration rate from pleth measured prospectively with either INVSENSOR00032 and/or INVSENSOR00033 devices against the respiration rate derived from the manual scoring of the capnography waveform in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Physical status of ASA I or II
* Must be able to read and communicate in English
* Has signed all necessary related documents, e.g. written informed consent, confidentiality agreement.
* Passed health assessment screening
* Negative pregnancy test for female subjects of child bearing potential.

Exclusion Criteria:

* Physical status of ASA III, IV, or V
* Subject has any medical condition which in the judgment of the investigator, renders them inappropriate for participation in this study
* Inability to tolerate sitting still or minimal movement for at least 30 minutes
* Positive pregnancy test for female subjects
* Refusal to take pregnancy test for women of child bearing potential
* Nursing female subjects
* Subjects wearing acrylic nails or subjects refusing to remove nail polish
* Subjects who have a nail deformity on the measurement finger
* Subjects who do not have adequate skin integrity on the measurement finger
* Excluded at the Principal Investigator's discretion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00032 and INVSENSOR00033 Test Group
Started | 27
Completed | 26
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00032 and INVSENSOR00033 Test Group
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 8
  Asian or Pacific Islander | 4
  Caucasian | 6
  Hispanic | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: RRp Arms of Sensor Accuracy
Description: Accuracy will be determined by comparing the noninvasive respiratory rate by pleth (RRp) measurement of the INVSENSOR00032 and/or INVSENSOR00033 to the respiratory rate reference (RRef) and calculating the arithmetic root mean square (Arms) value. In order to obtain the Arms value, the RR measurement from the reference is subtracted from the INVSENSOR00032 and/or INVSENSOR00033 RRp measurement for a number of samples. The average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms value.
Time Frame: 1-5 hours
Measure: Number; unit: respiration per minute (RPM)
Arm/Group | INVSENSOR00032 and INVSENSOR00033 Test Group
Number analyzed (Participants) | 26
respiration per minute (RPM) | 2.1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study (13 days).
Arm/Group | INVSENSOR00032 and INVSENSOR00033 Test Group
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT03897179/Prot_SAP_000.pdf